CLINICAL TRIAL: NCT03781882
Title: Local Injection of Autologous Platelet Rich Plasma During Repair of Disrupted Surgical Wounds at Obstetrics and Gynecology Department: A Randomized Controlled Study
Brief Title: Local Injection of PRP During Repair of Disrupted Surgical Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman S Dawood, MD, Lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRP surgical wounds
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Role of Platelet Rich Plasma in Wound Healing
Keywords: Platelet rich plasma; disrupted wounds; Obstetrics and Gynecology

STUDY DESIGN:
Intervention Model Description: All cases with disrupted surgical wounds admitted at Obstetrics and Gynecology departments
Who Masked: Participant
Masking Description: Patients were not allowed to know allocations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): All patients in this group will be manged as usual with infiltration of platelet rich plasma in thee wound edges during closure of the wounds
  Interventions: Procedure: Platelet rich plasma infiltration in the wound edges
- Control group (Active Comparator): All patients in this group will be managed by repair of wounds without infiltration of platelet rich plasma
  Interventions: Procedure: Closure of wound without platelet rich plasma infiltration

INTERVENTIONS:
Procedure: Platelet rich plasma infiltration in the wound edges — platelet rich plasma will be injected in the wound edges
  Arms: Intervention group
Procedure: Closure of wound without platelet rich plasma infiltration — No infiltration of platelet rich plasma is done
  Arms: Control group

SUMMARY:
Patients with disrupted wounds will either managed as usual or managed by Platelet rich plasma local infiltration in the wound edges

DETAILED DESCRIPTION:
The patients with disrupted surgical wounds will be cleansed, debrided and closed with infiltration of platelet rich plasma in one group and the other group will be closed without infiltration of Platelet rich plasma

ELIGIBILITY:
Inclusion Criteria:

* Disrupted surgical wounds after cesarean sections and other gynecological operations
* Body mass index 18-25
* Hemoglobin > 10.5gm/dl
* Albumin >3.5gm/dl

Exclusion Criteria:

* Medical disorders asDiabetes mellitus (DM), Liver disease or systemic lupus erythymatosus (SLE)
* Patient on corticosteriod therapy
* Thrombocytopenia
* Coagulation disorders

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Complete wound healing | 30 days
  time needed for complete wound closure
Duration of hospital stay | 30 days
  Time during which patient is admitted

SECONDARY OUTCOMES:
Failure of complete wound healing | 30 days
  No complete closure
Need fo tertiary suture | 30 days
  need to re-operate the case again

CONTACTS AND LOCATIONS:
Locations (1):
- Ayman Shehata Dawood, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
We will share unidentified data
Supporting Information: Study Protocol
Time Frame: 30 days